CLINICAL TRIAL: NCT06228898
Title: Does the Hematological Inflammatory Parameters Differ When Glycemic Control is Achieved in Patients With Type 2 Diabetes
Brief Title: Changes in Hematological Parameters With Glycemia Control in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: hematological parameters-T2D
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Poorly Controlled Diabetes Mellitus
Keywords: type 2 diabetes; glycemic control; neutrophils; neutrophil/lymphocyte ratio; lymphocyte/monocyte ratio; platelet/lymphocyte ratio; monocytes/HDL-cholesterol ratio; platelets/HDL ratio
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with type 2 diabetes with improved HbA1c: Participants with type 2 diabetes with a reduction in HbA1c ranging from 5% to 11.6% in three months time (n=56)
- patients with type 2 diabetes with a better HbA1c: Group 2 comprised individuals with type 2 diabetes who exhibited a decline in HbA1c levels ranging from 2.8% to 4.9% in three months time (n=56).
- patients with type 2 diabetes with little or no HbA1c change: Group 3 comprised 58 participants who exhibited a decrease in HbA1c levels ranging from 2.7% to 0%, in addition to an increase ranging from 0.1% to 3.4%.

SUMMARY:
There is a systemic low-grade chronic inflammation in diabetes, and research suggests that this inflammation plays a vital role in the development of diabetic complications. Macrovascular complications, which are associated with atherosclerosis, are recognized as a chronic inflammatory disease. In this study, the aim was to evaluate the potential alteration in hematologic inflammatory markers among patients with poorly controlled type 2 diabetes subsequent to the enhancement of diabetes management.

DETAILED DESCRIPTION:
Patients who were referred to the Diabetes Outpatient Clinics and had HbA1c levels equal to or greater than 10% were enrolled in this study. Detailed medical histories, comorbidities and medication usage (including both regular and new prescriptions), adherence to dietary recommendations, and occurence of recent infections were collected. Additionally, the patients' biochemical and hematological data were collected. After a three-month period, follow-up interviews with the same patients were conducted to inquire about any changes in medication usage, experienced illnesses, and hospital admissions. Based on the changes in HbA1c levels during this three-month period, the patients were divided into three equal groups. The baseline and third-month leukocyte counts, neutrophil counts, lymphocyte counts, and platelet counts for these groups were recorded. Furthermore, the neutrophil/lymphocyte ratio, lymphocyte/monocyte ratio, platelet/lymphocyte ratio, monocytes/HDL-cholesterol ratio, and platelets/HDL ratio for each group were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* having type 2 diabetes
* giving consent to the study
* HbA1c level >=10 %

Exclusion Criteria:

* presence of acute infection
* presence of other diseases that can cause inflammation
* hematological diseases
* acute metabolic decompensation
* not being able to come to follow-ups
* presence of non-thyroid endocrine disease
* application of oncologic treatment
* leukocyte count >12 000

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with poorly controlled type 2 diabetes, defined by an HbA1c level of >=10%, who attended diabetes outpatient clinics between January 2022 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
changes in hematologic inflammatory markers with glycemic control | three months
  to evaluate the potential alteration in hematologic inflammatory markers among patients with poorly controlled type 2 diabetes subsequent to the enhancement of diabetes management.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, MD, Principal Investigator — Goztepe Training and Research Hospital
Locations (1):
- Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No